CLINICAL TRIAL: NCT04301011
Title: A Phase 1/2a, Multicenter, Open-label Trial of TBio-6517, an Oncolytic Vaccinia Virus, Administered Alone and in Combination With Pembrolizumab, in Patients With Advanced Solid Tumors
Brief Title: Study of TBio-6517 Given Alone or in Combination With Pembrolizumab in Solid Tumors
Acronym: RAPTOR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Turnstone Biologics, Corp. (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBio-6517-ITu-001
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor; Microsatellite Stable Colorectal Cancer; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Cervical Cancer; Melanoma (Skin); Cutaneous Squamous Cell Carcinoma; Mesothelioma; Renal Cell Carcinoma; Oropharynx Cancer
Keywords: Renal Cell; CRC; MSS-CRC; Oncolytic Virus; Intratumoral injection; HPV cancer; cervical cancer; mesothelioma; melanoma; skin cancer; oropharyngeal
MeSH Terms: conditions — Uterine Cervical Neoplasms; Melanoma; Mesothelioma; Carcinoma, Renal Cell; Oropharyngeal Neoplasms; Skin Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm A: TBio-6517 alone (Experimental): Dose escalation of TBio-6517 alone administered by direct injection into tumor(s) x 4. Booster injections of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517
- Arm B: TBio-6517 and Pembrolizumab (Experimental): Dose escalation of TBio-6517 administered in combination with pembrolizumab. TBio-6517 will be directly injected into tumor(s) x 4. Booster injections of TBio-6517 are permitted for up to 24 months. Pembrolizumab will be administered beginning at Day 9 via intravenous (IV) infusion every 3 weeks for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab
- TBio-6517 and Pembrolizumab in MSS-CRC (Experimental): Doses of TBio-6517 will be administered by direct injection into tumor(s) x 4 in combination with pembrolizumab beginning at Day 9 given every 3 weeks for up to 24 months in patients with microsatellite stable colorectal carcinoma (MSS-CRC). Booster injections of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab
- TBio-6517 and Pembrolizumab in cutaneous melanoma (Experimental): Doses of TBio-6517 will be administered by direct injection into tumor(s) x 4 in combination with pembrolizumab beginning at Day 9 given every 3 weeks for up to 24 months in patients with malignant melanoma of the skin. Booster injections of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab
- TBio-6517 and Pembrolizumab in cutaneous squamous cell carcinoma of the skin (Experimental): Doses of TBio-6517 will be administered by direct injection into tumor(s) x 4 in combination with pembrolizumab beginning at Day 8 given every 3 weeks for up to 24 months in patients with cSCC. Booster injections of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab
- TBio-6517 and Pembrolizumab in HPV positive head and neck cancer (Experimental): Doses of TBio-6517 will be administered by direct injection into tumor(s) x 4 in combination with pembrolizumab beginning at Day 9 given every 3 weeks for up to 24 months in patients with HPV associated oropharyngeal cancer. Booster injections of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab
- Arm C: TBio-6517 intravenous (Experimental): Dose escalation of TBio-6517 alone administered by intravenous infusion x 4. Booster infusions of TBio-6517 are permitted for up to 24 months.
  Interventions: Biological: TBio-6517
- Arm D: TBio-6517 intravenous and Pembrolizumab (Experimental): Dose escalation of TBio-6517 administered in combination with pembrolizumab. Dose escalation of TBio-6517 alone administered by intravenous infusion x 4. Booster infusions of TBio-6517 are permitted for up to 24 months. Pembrolizumab will be administered beginning at Day 9 via intravenous (IV) infusion every 3 weeks for up to 24 months.
  Interventions: Biological: TBio-6517; Biological: Pembrolizumab

INTERVENTIONS:
Biological: TBio-6517 — Engineered Oncolytic Vaccinia Virus
  Other Names: RIVAL-01
Biological: Pembrolizumab — Immune checkpoint inhibitor.
  Other Names: Keytruda
  Arms: Arm B: TBio-6517 and Pembrolizumab; Arm D: TBio-6517 intravenous and Pembrolizumab; TBio-6517 and Pembrolizumab in HPV positive head and neck cancer; TBio-6517 and Pembrolizumab in MSS-CRC; TBio-6517 and Pembrolizumab in cutaneous melanoma; TBio-6517 and Pembrolizumab in cutaneous squamous cell carcinoma of the skin

SUMMARY:
To determine the recommended Phase 2 dose (RP2D) of TBio-6517 when administered by direct injection into tumor(s) or intravenously and when combined with pembrolizumab in patients with solid tumors (RIVAL-01).

DETAILED DESCRIPTION:
This is a Phase 1/2a dose escalation study with TBio-6517 administered by direct injection into tumor(s) or by intravenous infusion. The Phase 1 portion has 4 arms; the first arm (Arm A) will determine the RP2D of TBio-6517 alone when directly injected into tumor(s), and the second arm (Arm B) will determine the RP2D of TBio-6517 when combined with pembrolizumab. The third and fourth arms will determine the RP2D of TBio-6517 when given intravenously alone and with pembrolizumab, respectively.

In the Phase 2a portion, the clinical benefit of TBio-6517 combined with pembrolizumab will be further explored in patients with Microsatellite Stable Colorectal Cancer (MSS-CRC), Cholangiocarcinoma (CCA), Cutaneous Melanoma, and Cutaneous Squamous Cell Carcinoma of the Skin (cSCC), as assessed by overall response rate (ORR) from central radiology review.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a histologically or pathologically documented, locally-advanced or metastatic solid tumor for which standard curative measures do not exist or are no longer effective
* Measurable disease as per RECIST 1.1 criteria
* At least one tumor amenable to safe ITu injections and biopsies
* ECOG performance status 0 or 1
* Demonstrate adequate organ function
* Must be willing to comply with all protocol procedures and adhere to post-treatment care instructions
* Additional Inclusion criteria exist

For patients in phase 2 only: Have a histologically or cytologically confirmed advanced (metastatic and/or unresectable) solid tumor listed below, that is incurable and for which prior standard treatment has failed:

1. Advanced (unresectable) or metastatic, intra or extra hepatic adenocarcinoma originating from the bile duct, CCA (Cohort 1) having progressed on at least 1 line of systemic therapy (including targeted therapy if eligible)
2. Locally advanced or metastatic cutaneous melanoma (Cohort 2) that has failed anti-PD-1 or anti-PDL1 therapy (+/- anti-CTLA-4 therapy) and if BRAF+, having failed a BRAF/ +/-MEK inhibitor
3. Locally advanced or metastatic cSCC (Cohort 3) that has not received systemic therapy (e.g., local resection or local topical therapy is permitted).
4. Locally advanced or metastatic MSS-CRC (Cohort 4) patients that have progressed on at least 2 prior lines of systemic therapy which should include irinotecan and oxaliplatin +/- targeted therapy if warranted.

Key Exclusion Criteria:

* Prior systemic therapy, including experimental, surgery or radiation therapy within 4 weeks and must have recovered from acute toxicity.
* Prior treatment with any oncolytic virus.
* Requires use of anti-platelet or anti-coagulant therapy that cannot be safely suspended for per protocol biopsies or intra-tumoral injections.
* CNS metastases and/or carcinomatous meningitis that have not been completely resected or completely irradiated.
* Prior history of myocarditis
* Symptomatic or asymptomatic cardiovascular disease
* Known HIV/AIDS, active HBV or HCV infection.
* Received immunosuppressive medication within 4 weeks. (>10mg/day prednisone)
* Known intolerance to anti-PD-1 or anti-PD-L1 antibody therapy
* Additional Exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events when TBio-6517 administered by direct injection into tumor(s) alone at each dose level | 25 months
  Percentage of patients with adverse events by grade as determined by NCI CTCAE v5.0
Incidence of adverse events when TBio-6517 administered by direct injection into tumor(s) when combined with pembrolizumab | 25 months
  Percentage of patients with adverse events by severity as determined by NCI CTCAE v5.0
Maximum tolerated dose (MTD) or Maximum feasible dose (MFD) and determination of the recommended Phase 2 dose (RP2D) of TBio-6517 alone and in combination with pembrolizumab. | 4 weeks
  The highest dose of TBio-6517 that can be administered where fewer than 2 patients have a dose-limiting safety event alone or when combined with pembrolizumab as assessed by NCI CTCAE v.5.0 during the Phase 1 dose escalation
Percentage of overall response rate (ORR) by RECIST 1.1 at the RP2D | 25 months
  Percentage of patients treated at the RP2D in combination with pembrolizumab with a partial response or complete response by RECIST 1.1 following central radiologist review
Percentage of overall response rate (ORR) by immunotherapy RECIST (iRECIST) at the RP2D | 25 months
  Percentage of patients treated at the RP2D with pembrolizumab with a partial response (PR) or complete response (CR) by iRECIST following central radiologist review

SECONDARY OUTCOMES:
Number and severity of adverse events at the RP2D | 25 months
  Number of patients with adverse events by severity and frequency as determined by NCI CTCAE v5.0
Median overall survival (OS) | 48 months
  Median overall survival in months in patients
Median Duration of Response (DoR) | 25 months
  Median duration of response in patients with a CR or PR
Proportion of patients with a response (ORR) | 25 months
  Percentage of patients in all arms with a CR or PR as assessed by the central radiologist using RECIST 1.1 and iRECIST
Median Disease Control Rate (DCR) | 25 months
  Median duration of response in patients with a CR, PR, or stable disease (SD)
Time to tumor progression (TTP) | 25 months
  Median time until patient disease progression (PD)
Median progression free survival | 25 months
  Median duration of progression free survival of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ines Verdon, MD, Study Director — Turnstone Biologics
Locations (11):
- United States (8):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center / UMHC, Miami, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Clinical Site 1007, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The Billings Clinic, Billings, Montana
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Ottawa Hospital and Research Institute (OHRI), Ottawa, Ontario, Canada
- South Korea (2):
  - National Cancer Center, Ilsandong
  - Seoul National University Hospital (SNUH), Junggu